CLINICAL TRIAL: NCT01556789
Title: Phase 1 Study of ONT-10, a Liposomal MUC1 Cancer Vaccine, in Patients With Solid Tumors
Brief Title: Phase 1 Study of ONT-10 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cascadian Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONT-10-001
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2015-09

CONDITIONS: Solid Tumors
Keywords: ONT-10; MUC1; Vaccine; Phase 1; Solid Tumors; Dose escalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ONT-10 Vaccine (Experimental): ONT-10 investigational agent
  Interventions: Biological: ONT-10

INTERVENTIONS:
Biological: ONT-10 — ONT-10 a liposomal synthetic glycolipopeptide antigen formulated with PET Lipid A adjuvant.

SUMMARY:
Open label, two part, Phase 1 dose escalation study to evaluate the safety and immunogenicity of repeat dose vaccination with ONT-10 in patients with previously treated Stage 3 or 4 solid tumors. Part 1 to evaluate escalating dose levels of ONT-10 administered subcutaneously every two weeks (Q2W) or weekly (QW) over 8 weeks. Part 2 evaluates the safety, immunogenicity, and potential anti-tumor activity of ONT-10 administered over 8 weeks at the Q2W and QW maximum tolerated does/recommended dose (MTD/RD) in cohorts of 15 patients each.

DETAILED DESCRIPTION:
This open label, two part, Phase 1 dose escalation study will evaluate the safety and immunogenicity of repeat dose vaccination with ONT-10 in patients with previously treated Stage 3 or 4 solid tumors with histologies that have been associated with expression of the MUC1 antigen as described in the medical literature. Part 1 will evaluate escalating dose levels of ONT-10 administered subcutaneously Q2W over 8 weeks (for a total of 4 doses) or QW over 8 weeks (for a total of 8 doses) to identify a MTD and/or RD for each dosing schedule, for further evaluation in Part 2 of the study. Part 2 will evaluate the safety, immunogenicity, and potential anti-tumor activity of ONT-10 administered over 8 weeks at the Q2W and QW MTD/RD in cohorts of 15 patients each.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 to 70 years of age at time of consent
2. Life expectancy of at least 6 months, in the opinion of the investigator
3. A) Have histologically confirmed breast, non-small cell lung, ovarian, colorectal, gastric, prostate, pancreatic, or renal cell cancer, or other tumor type as approved by the study medical monitor (Part 1) B) Have histologically confirmed breast or ovarian carcinoma (Part 2)
4. Have evidence of persistent, recurrent, or progressive disease after at least one course of systemic therapy for locally advanced or metastatic disease, including chemotherapy, targeted therapy, or immunotherapy
5. Clinical stage 3 or 4 disease
6. ECOG 0 or 1
7. Adequate baseline hematological parameters as defined by white blood cell count (WBC) ≥ 3.5 x 103/uL, lymphocyte count ≥ 1.0 x 103/uL, platelet count ≥ 100 x 103/uL, and hemoglobin ≥ 9 g/dL
8. Have renal and hepatic function laboratory test results not to exceed 1.5 X upper limit of normal (ULN)
9. If female of child bearing potential, have a negative pregnancy test at screening
10. If fertile male or female of child-bearing potential, agree to consistently use a highly effective method of birth control (including birth control pills, barrier device, or intrauterine device) from the time of consent through 3 months following the last dose of study drug.
11. Be able and willing to sign informed consent document that has been approved by an institutional review board or independent ethics committee (IRB/IEC)

Exclusion Criteria:

1. Has medical, social, or psychosocial factors that, in the opinion of the investigator, could impact safety or compliance with study procedures
2. Is pregnant, breastfeeding, or planning a pregnancy
3. Has received treatment with any systemic chemotherapy, radiation, or experimental agent within 4 weeks of study drug dosing
4. Has untreated or uncontrolled central nervous system (CNS) metastases, including patients who require glucocorticoid therapy for CNS metastases.
5. Has a known history of autoimmune disease, arteritis, or vasculitis, including, but not limited to: lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease (including ulcerative colitis and Crohn's disease), Grave's disease, Hashimoto's thyroiditis, Wegener's granulomatosis, temporal arteritis, and polyarteritis nodosa
6. Has a recognized immunodeficiency disease, including cellular immunodeficiencies, hypogammaglobulinemia, or dysgammaglobulinemia; and/or other hereditary or congenital immunodeficiencies
7. Has any preexisting medical condition requiring chronic steroid or immunosuppressive therapy (corticosteroids for COPD or topical steroids are allowed)
8. Known to be positive for HIV, hepatitis B, or hepatitis C
9. Administration of any other vaccine ≤ 4 weeks prior to study enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety | 20 weeks
  Assessment of adverse events and laboratory abnormalities

SECONDARY OUTCOMES:
Immunogenicity | 20 weeks
  Assessments to include evaluation of humoral and cellular immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Hausman, MD, Study Chair — Cascadian Therapeutics Inc.
Locations (3):
- United States (3):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington